CLINICAL TRIAL: NCT05962788
Title: An Open-Label Extension Study to Assess the Long-Term Safety and Efficacy of Voclosporin in Adolescent and Pediatric Subjects With Lupus Nephritis
Brief Title: Long-Term Voclosporin Treatment in Adolescent and Pediatric Subjects With Lupus Nephritis
Acronym: VOCAL-EXT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB recommendation
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUR-VCS-2020-04
Record Dates: First submitted 2023-06-21; First posted 2023-07-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Adolescent Lupus Nephritis; Pediatric Lupus Nephritis
Keywords: voclosporin; lupus nephritis; calcineurin inhibitors; adolescents; pediatrics
MeSH Terms: conditions — Lupus Nephritis | interventions — voclosporin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label (Experimental): All subjects will receive open label voclosporin initially at the same number of capsules as assigned at Week 24 (End of Study Visit) in AUR-VCS-2020-03 (VOCAL ; NCT05288855). At the Investigator's discretion and after consultation with the Medical Monitor, dose titration up or down in the study will be permitted up to the maximum dose that was studied in AUR-VCS-2020-03.
  Interventions: Drug: voclosporin

INTERVENTIONS:
Drug: voclosporin — Subjects will receive 2 capsules (15.8 mg) BID (twice daily), 3 capsules (23.7 mg) BID of voclosporin in addition to standard of care with mycophenolate mofetil (MMF) and steroids.

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of voclosporin for up to an additional 12 months following completion of treatment in the AUR-VCS-2020-03 study (VOCAL) in adolescent and pediatric subjects with lupus nephritis.

DETAILED DESCRIPTION:
This is a 12 month, prospective, multi-center, long-term, open-label extension study of voclosporin in addition to background standard of care with mycophenolate mofetil (MMF) and oral steroids.

Subjects completing participation and treatment with study drug (voclosporin/placebo) of the VOCAL Study (AUR-VCS-2020-03 ; NCT05288855) and meeting all eligibility criteria will receive open-label treatment with voclosporin for approximately 12 months giving a total study treatment duration of 18 months from the start of VOCAL.

All subjects will continue to receive background therapy of MMF and oral corticosteroids starting at the same dose as at completion of the VOCAL study. When clinically indicated, subjects are permitted to be titrated off oral corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from parent/guardian before any study-specific procedures are performed, if applicable per local regulations.
* Age-appropriate assent or informed consent from subject before any study-specific procedures are performed.
* Subjects who have completed 24 weeks of treatment with study drug (voclosporin/placebo) in the VOCAL study. Subjects who had a temporary interruption and were able to successfully re-start study drug will be allowed to enroll after Medical Monitor approval.
* In the opinion of the Investigator subject requires continued immunosuppressive therapy.
* Subject is willing to continue to take oral MMF for the duration of the study.

Exclusion Criteria:

* Currently taking or known need for any of the following medications during the study:

  * Cholestyramine or other drugs that may interfere with enterohepatic recirculation of MMF
  * Calcineurin inhibitors (CNIs) (e.g., cyclosporin and tacrolimus)
  * Strong CYP3A4/5 inhibitors and inducers (e.g., ketoconazole, rifampin, itraconazole, clarithromycin)
* Currently requiring renal dialysis (hemodialysis or peritoneal dialysis) or expected to require dialysis during the study period.
* A planned kidney transplant within study treatment period.
* Subjects with any medical condition which in the Investigator's judgement may be associated with increased risk to the subject or may interfere with study assessments or outcomes

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAE) | Per protocol from VOCAL-EXT Study Start to Study Completion plus a 30-day follow-up period
  Incidence (subject counts and event counts) of TEAEs summarized by System Organ Class and Preferred Terms using MedDRA

SECONDARY OUTCOMES:
Renal Response | Per protocol from Study Start to Study Completion plus a 30-day follow-up period
  Proportion of subjects with renal response at Month 12 and 18, defined based on the following parameters:
  * urine protein creatinine ratio (UPCR) of ≤0.5 mg/mg, and
  * estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73 m2 or no confirmed decrease from baseline in eGFR of >20%, and
  * Received no rescue medication for lupus nephritis, and
  * Did not receive >10 mg/day prednisone for ≥3 consecutive days or for ≥7 days in total prior to the renal response assessment
Urine Protein Creatinine Ratio (UPCR) | Month 12 (VOCAL Study Completion/VOCAL-EXT Study Start) and Month 18 (VOCAL-EXT Study Completion)
  Proportion of subjects with UPCR of ≤0.7 mg/mg
Partial Renal Response | Month 12 (VOCAL Study Completion/VOCAL-EXT Study Start) and Month 18 (VOCAL-EXT Study Completion)
  Proportion of subjects in partial renal response as defined by ≥50% reduction from VOCAL baseline in UPCR

CONTACTS AND LOCATIONS:
Locations (6):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States
- Clinica de la Costa S.A.S, Barranquilla, Atlántico, Colombia
- Yokohama City University Hospital, Yokohama, Kanagawa, Japan
- Mexico (2):
  - Centro de Especialidades Medicas del Sureste, Mérida, Yucatán
  - Hospital Infantil de México Federico Gómez, Mexico City
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No